CLINICAL TRIAL: NCT01235325
Title: The Effect of Vitamin K Supplementation on Bone Health Indices in Adult Crohn's Disease
Brief Title: The Effect of Vitamin K Supplementation on Bone Health in Adult Crohn's Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Health Research Board, Ireland (Other)
Responsible Party: Professor Kevin D. Cashman, University College Cork, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRB RP/2006/38
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Supplementation; Bone Health; Crohn's Disease
Keywords: vitamin K; supplementation; bone health indices; adult; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Vitamin K 1

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo oil capsule (Placebo Comparator): Banner Pharmacaps Europe
  Interventions: Dietary Supplement: placebo
- phylloquinone (1000 mcg) (Experimental): Banner Pharmacaps Europe
  Interventions: Dietary Supplement: phylloquinone (vitamin K1)

INTERVENTIONS:
Dietary Supplement: phylloquinone (vitamin K1) — 1000 mcg phylloquinone (vitamin K1) once daily for 12 months
  Other Names: Banner Pharmacaps Europe
  Arms: phylloquinone (1000 mcg)
Dietary Supplement: placebo — placebo oil capsule
  Other Names: Banner Pharmacaps Europe
  Arms: Placebo oil capsule

SUMMARY:
To assess the impact of a 12 month vitamin K supplementation intervention on bone health in adult Crohn's disease patients

DETAILED DESCRIPTION:
To assess the impact of 12 months of vitamin K1 supplementation (plus vitamin D and calcium supplementation to avoid deficiency of these problematic nutrients) at a level which leads to dramatically (i.e greater than 70%) reduced levels of undercarboxylated osteocalcin - a functional marker of vitamin K status, on vitamin K status, the rate of bone formation and bone resorption, using biochemical markers of bone turnover, and bone mineral density in adult patients with longstanding Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* long-standing Crohn's disease - disease diagnosis > 5 years
* in clinical remission at baseline - Harvey-Bradshaw score (< 5)
* aged between 18-70 years

Exclusion Criteria:

* use of steroid medications to treat disease or flare up
* use of blood thinning medications (warfarin, heparin, asprin, dicoumarol derivatives) which may influence vitamin K metabolism
* use of bisphosphonates, calcitonin medications (to treat osteoporosis)
* use of experimental drugs (in the last 30 days) or inclusion in another intervention trial
* bone mineral density < -2.5 (indicative of osteoporosis) or previous diagnosis of osteoporosis
* use of vitamin/mineral/fish liver oil dietary supplements
* use of other alternative supplements (i.e herbal)
* if the patient is under 18 or over 70 years of age
* presence of a significant acute or chronic coexisting illness (cardiovascular, immunological or a condition which in the investigator's judgement, contraindicates involvement in the study)
* presence of malignant or any concomitant end-stage organ disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
% Undercarboxylated osteocalcin | 12 months
  Measurement of carboxylated and undercarboxylated osteocalcin (expressed as %) as a senstive functional marker of vitamin K status.

SECONDARY OUTCOMES:
25-Hydroxy vitamin D (25OHD) | 12 months
  Measurement of serum 25-Hydroxy vitamin D as status measure
Intact Parathyroid hormone (iPTH) | 12 months
  Measurement of intact parathyroid hormone to determine hyperparathyroidism, hypercalcemia, vitamin D deficiency
Urinary creatinine | 12 months
  For standardisation of urinary NTx measurement
Serum phylloquinone | 12 months
  Determination of serum phylloquinone by HPLC
Biochemical markers of bone turnover (BAP, CTx, NTx) | 12 months
  Use of biochemical markers of bone turnover to assess the effect of supplementation on bone health.
Bone mineral density (BMD) | 12 month
  Measurement of bone mineral density (BMD) by iDEXA
Food Frequency Questionnaire (FFQ) for habitual vitamin K, vitamin D and calcium intakes | cross-sectional (baseline only)
  Food frequency questionnaire (FFQ) to estimate habitual vitamin K (vitamin D and calcium) status, cross-sectionally at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Cashman, Professor, Principal Investigator — University College Cork, Ireland; Fergus Shanahan, Professor, Study Director — University College Cork, Ireland
Locations (1):
- Clinical Investigations Unit, Cork University Hospital, Wilton, Cork, Co. Cork, Ireland